CLINICAL TRIAL: NCT05706389
Title: Does Alpha-ketoglutarate Supplementation Lower BiologicaL agE in Middle- Aged Adults?
Acronym: ABLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Agency for Science, Technology and Research (Other); AMILI Pte. Ltd. (Unknown)
Responsible Party: Principal Investigator, Andrea Maier, Oon Chiew Seng Professor in Medicine, Healthy Ageing and Dementia Research, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NUS-IRB-2021-946
Record Dates: First submitted 2022-12-25; First posted 2023-01-31 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Aging
Keywords: Aging; Geroscience; Alpha-Ketoglutarate; DNA methylation; Healthspan; epigenetic aging clock

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-controlled longitudinal interventional study on middle-aged participants
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ca-AKG (Experimental): Pill format, 500mg/pill, half of daily dose
  Interventions: Dietary Supplement: Ca-AKG
- Placebo (Placebo Comparator): Pill format, indistinguishable from active pill
  Interventions: Dietary Supplement: Ca-AKG

INTERVENTIONS:
Dietary Supplement: Ca-AKG — Eligible participants will be randomised to receive Ca-AKG or Placebo for 6 months.

SUMMARY:
Geroscience is an emerging interdisciplinary field of study in gerontological sciences. With emphasis on understanding the mechanistic drivers of aging, it seeks translational approaches that could eventually be applied to improve human healthspan and delay age-associated chronic diseases. Contrary to popular opinion that aging is irreversible, advances in geroscience research have demonstrated that aging is modifiable and inhibiting or activating specific molecular pathways can improve healthspan and extend lifespan in model organisms. Advocates of geroscience take the view that age-related chronic diseases are best treated by slowing the aging process, rather than using the prevailing disease-centric approach of addressing each disease alone. Thus, the concept is that biological aging, rather than chronological aging, is amenable to intervention.

In this regard, geroscientists are at the forefront of longevity medicine in rigorously testing novel supplements, drugs and other prophylactics that can enhance healthspan. Some of these interventions involve repurposing existing drugs such as rapamycin, a well-known immunosuppressant, at different dosing regimens to specifically target biological hallmarks of aging.

This study will investigate the effects of alpha-ketoglutarate (AKG), an endogenous metabolite, on biomarkers of aging in middle-aged residents of Singapore.

DETAILED DESCRIPTION:
Recent growing understanding on mechanisms of aging as gradual changes in body systems through several cellular and molecular levels has raised research interests in the biology of aging. There are seven established overlapping processes of aging: oxidative stress, macromolecular damage, epigenetic changes, abnormal metabolism, impaired proteostasis, decline in stem cell functions and inflammation. These overlapping changes over the lifetime affect the onset of age-related diseases and possibly the aging process itself. However, lifestyle and pharmacologic interventions can modify the deterioration of aging pathways. AKG is a generally regarded as safe (GRAS) micronutrient and has shown great potential in extending healthspan. Here, we aim to study the role of AKG in the modulation of aging.

The aim is to evaluate the anti-aging function of AKG and determine whether AKG can modulate biological pathways of aging in middle-aged adults in Singapore. Our hypothesis is that AKG will affect DNA methylation which will be associated with the change in blood biomarkers of aging and change in physiological function. It allows us to study the longitudinal effects of AKG on clinical and biological outcomes.

This is a 6-month double-blinded, placebo-controlled longitudinal interventional study on middle-aged participants to study the effect of AKG on biomarkers of aging, with another 3 months of post-intervention follow-up. The total duration of participation in this study is 9 months.

The rationale for this study design is to study the long-term effect of 1 g AKG in middle-aged adults. Our study design of 6 months of intervention (1 g AKG vs placebo) will allow us to understand the effect of AKG treatment on DNA methylation, and another 3 months of post-intervention follow-up will help us understand if there is any long-term effect of AKG. In order to minimize recruitment bias, our study design is double-blinded.

ELIGIBILITY:
Inclusion Criteria:

* participants whose biological age (as measured by blood DNA methylation) is greater than their chronological age

Exclusion Criteria:

* pregnant women
* more than ONE of the following chronic medical conditions (based on the medical history and during screening), they are NOT eligible to participate in the study:

  1. Waist circumference more than or equal to 90 cm for males or more than or equal to 80 cm for females
  2. Fasting triglycerides more than or equal to 1.7 mmol/l
  3. High-density lipoprotein less than 1.0 mmol/l in men or less than 1.3 mmol/l in women
  4. Blood pressure more than or equal to 130/85 mmHg or use of antihypertensive medication
  5. Fasting glucose more than or equal to 6.0 mmol/l
  6. Osteopenia
  7. Mild Osteoarthritis not interfering in daily activities
  8. Fatty liver
* Participants will NOT be recruited if they fall in the following categories:

  1. Pre-existing, or history of major CVD (coronary artery disease, heart failure, stroke, peripheral vascular disease, pulmonary hypertension), severe/uncontrolled hypertension (under 3 or more than 3 prescribed medications), rheumatic heart disease, congenital heart disease, deep vein thrombosis, pulmonary embolism
  2. Type 1 diabetes and Type 2 diabetes under oral metformin or insulin therapy and with diabetic complications such as diabetic retinopathy, diabetic nephropathy
  3. Active cancer or treatment of cancer in the last 3 years
  4. Chronic obstructive pulmonary disease (COPD), severe asthma (taking daily medications)
  5. Pregnant women will not be recruited into this study because of the safety issues associated with X-ray irradiation during DXA scan
  6. Potential female participants who plan on pregnancy within the next 9 months of study period
  7. Multiple sclerosis and autoimmune/immune deficiency diseases such as Rheumatic arthritis, HIV, Crohn's disease
  8. Recent history of sepsis or infection (within 3 months of in-patient hospitalization)
  9. Any psychiatric disease or neurodegenerative diseases such as Alzheimer's Disease, Parkinson's Disease, Lewy body dementia, and any eating disorders
  10. Any metal implants in the body
  11. Hepatitis and Liver cirrhosis (independent of severity)
  12. Severe kidney disease (GFR less than 30 ml/min/1.73 m2)
  13. Skin disease (on oral or systemic medication for immune system)
  14. Subjects receiving any other similar investigational product within 60 days or 5 halflives before the screening, whichever that is longer
  15. Any serious medical illness which in the PI's judgment may jeopardize the subject by his or her participation in this study or may hamper his or her ability to perform and complete procedures required in the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in blood DNA methylation status, years | from baseline to end of intervention (6 months)
  DNA methylation aging clock

SECONDARY OUTCOMES:
Complete blood count | from baseline to end of intervention (6 months)
  comparison of blood count at baseline and 6 months
Carotid-femoral Pulse Wave Velocity change | from baseline to end of intervention (6 months)
  comparison of PWV at baseline and 6 months
Central Blood pressure change | from baseline to end of intervention (6 months)
  comparison of Central Blood pressure at baseline and 6 months
Body Mass Index (BMI) change | from baseline to end of intervention (6 months)
  comparison of BMI at baseline and 6 months
Brachial Blood pressure change | from baseline to end of intervention (6 months)
  comparison of Brachial Blood pressure at baseline and 6 months
Waist/hip ratio change | from baseline to end of intervention (6 months)
  comparison of Waist/hip ratio at baseline and 6 months
Bone Mineral Density, g/cm2 change | from baseline to end of intervention (6 months)
  comparison of Bone Mineral Density at baseline and 6 months
Fat-free mass, change (kg) | from baseline to end of intervention (6 months)
  comparison of fat-free mass at baseline and 6 months
Fat mass, change (kg) | from baseline to end of intervention (6 months)
  comparison of fat mass at baseline and 6 months
Handgrip strength change (kg) | from baseline to end of intervention (6 months)
  comparison of handgrip strength at baseline and 6 months
8-RM leg extension change (kg) | from baseline to end of intervention (6 months)
  comparison of 8RM leg extension at baseline and 6 months
Cardiopulmonary exercise test (CPET): Change in Volume of Oxygen consumption (V̇O2), L/min | from baseline to end of intervention (6 months)
  comparison of VO2 during CPET at baseline and 6 months
Cardiopulmonary exercise test (CPET): Change in Volume of Oxygen consumption per kg body weight (V̇O2/kg), L/min/kg | from baseline to end of intervention (6 months)
  comparison of VO2/kg during CPET at baseline and 6 months
Cardiopulmonary exercise test (CPET): change in lactate | from baseline to end of intervention (6 months)
  comparison of lactate levels during CPET at baseline and 6 months
Cardiopulmonary exercise test (CPET): change in heart rate | from baseline to end of intervention (6 months)
  comparison of heart rate levels during CPET at baseline and 6 months
Cardiopulmonary exercise test (CPET): aerobic and anaerobic threshold change | from baseline to end of intervention (6 months)
  comparison of aerobic and anaerobic threshold levels during CPET at baseline and 6 months
Cardiopulmonary exercise test (CPET): excess post-exercise oxygen consumption change | from baseline to end of intervention (6 months)
  comparison of excess post-exercise oxygen consumption levels during CPET at baseline and 6 months
Change in Skin autofluorescence, au | from baseline to end of intervention (6 months)
  comparison of skin autofluorescence levels at baseline and 6 months
Change in Quality-of-Life questionnaires (SF-36 questionnaires) | from baseline to end of intervention (6 months)
  comparison of Quality-of-life at baseline and 6 months
Change in Quality-of-Life questionnaires (EuroQoL-5D-5L) | from baseline to end of intervention (6 months)
  comparison of Quality-of-life at baseline and 6 months
Change in Sleep (modified Pittsburgh sleep quality Questionnaire ) | from baseline to end of intervention (6 months)
  comparison of sleep at baseline and 6 months
Change in Sleep (Satisfaction, Alertness, Timing, Efficiency and Duration (SATED) Questionnaire ) | from baseline to end of intervention (6 months)
  comparison of sleep at baseline and 6 months
Change in Global preferences survey (GPS) | from baseline to end of intervention (6 months)
  comparison of global preferences (GPS) at baseline and 6 months
AKG, glutamate, glutamine concentrations in serum | from baseline to end of intervention (6 months)
  Metabolites in serum change
Change in Immune parameters (Complete Blood Count) | from baseline to end of intervention (6 months)
  Immune parameters change
Change in Immune parameters (inflammatory parameters in serum, mg/dL) | from baseline to end of intervention (6 months)
  Immune parameters change
Change in Clinical Blood parameters: Renal function, mg/dL | from baseline to end of intervention (6 months)
  Clinical Blood parameters change
Change in Clinical Blood parameters: Lipid profile test, mmol/L | from baseline to end of intervention (6 months)
  Clinical Blood parameters change
Change in Clinical Blood parameters: Glucose, mg/dL | from baseline to end of intervention (6 months)
  Clinical Blood parameters change
Change in Clinical Blood parameters: insulin, mg/dL | from baseline to end of intervention (6 months)
  Clinical Blood parameters change
Change in Clinical Blood parameters: HbA1C, mmol/mol | from baseline to end of intervention (6 months)
  Clinical Blood parameters change
Change in Clinical Blood parameters: Metabolites, mmol/l | from baseline to end of intervention (6 months)
  Clinical Blood parameters change
Change in Cognitive function test by Montreal Cognitive Assessment (MoCA) | from baseline to end of intervention (6 months)
  Cognitive function change
Change in saliva DNA methylation status, years | from baseline to end of intervention (6 months)
  DNA methylation aging clock

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Healthy Longevity, Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No